CLINICAL TRIAL: NCT06372834
Title: Efficacy of Adjuvant Accelerated Prolonged Intermittent Theta Burst Stimulation for Reducing Suicidal Ideation in Therapy-resistant Depressed Patients: A Randomized, Sham-controlled Trial
Brief Title: Adjuvant Accelerated piTBS for Reducing Suicidal Ideation in TRD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Hsin-An Chang, MD, Attending Psychiatrist, Department of Psychiatry, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B202205178
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder; Treatment-Resistant Depression; Suicide Ideations
Keywords: Major Depressive Disorder; Treatment-Resistant Depression; Dorsolateral prefrontal cortex; rTMS; piTBS
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- piTBS (active, N=50) (Experimental): The piTBS sessions will be delivered using the Magstim Rapid2 stimulator (Magstim Company, Ltd, Whitland, Wales, UK, SA340HR) with a 70-mm air-cooled figure-eight coil (Magstim D70 Air film coil). The piTBS protocol consists of 3-pulse 50-Hz bursts given every 200 ms (at 5 Hz) for 2 s at 8-s intervals for 60 cycles. A 2-s train of piTBS will be repeated every 10 s for a total of 1800 pulses per session. The intensity of stimulation will be set at 90% resting motor threshold (RMT), as measured from the right first dorsal interosseous muscle by a handheld 700-mm figure-of-eight coil (Magstim D70 alpha coil). The Beam F3 method will be used for coil positioning to target the left dorsolateral prefrontal cortex. The piTBS protocol will be scheduled for 3 sessions per working day for 2 weeks (i.e., a total of 30 sessions over 2 weeks). Three sessions of the piTBS per day will be separated by at least 60 mins.
  Interventions: Device: piTBS being delivered using the Magstim Rapid2 stimulator
- piTBS (sham, N=50) (Sham Comparator): The patients in the sham piTBS condition will receive the same piTBS regimen and exact positioning of the coil, but stimulations will be delivered using a commercial identical-looking figure-8 sham coil (Magstim D70 Air film sham coil) that can produce a similar sound and sensations but induce neither magnetic pulses nor current in the cortex.
  Interventions: Device: piTBS being delivered using the Magstim Rapid2 stimulator

INTERVENTIONS:
Device: piTBS being delivered using the Magstim Rapid2 stimulator — Magstim Rapid2 stimulator (Magstim Company, Ltd, Whitland, Wales, UK, SA340HR). See detail in arm/group descriptions regarding the intervention.

SUMMARY:
In this double-blind, randomized, sham-controlled trial, the investigators aimed to examine the effect of accelerated piTBS on suicide risk in a group of treatment-resistant patients with MDD (i.e., TRD), using an extensive suicide assessment scale the primary outcome. The investigators hypothesized that this intensified treatment protocol would be safe in TRD patients with suicide ideations and would result in significant decreases in suicide risk in the active treatment condition as compared to the sham condition.

DETAILED DESCRIPTION:
Less than half of patients with major depressive disorder (MDD) remit after first-line therapy (i.e., pharmacotherapy and/or psychotherapy). A progressively smaller proportion of patients remit with each subsequent medication trial, and a remission rate of only 10-15% after a fourth antidepressant trial. Patients with MDD are considered to have a treatment-resistant depression (TRD) whey they do not achieve response to first-line antidepressants. Repetitive Transcranial Magnetic Stimulation (rTMS) applied over the DLPFC for modulating brain activity and network connectivity has well-documented positive effects on major depressive disorder (MDD), especially TRD. rTMS research in treating MDD has shown a dose-response relationship and more recently, studies have shown a trend towards administering more stimuli over a shorter period of time and at higher frequencies leading to accelerated protocols. An optimized rTMS parameter called intermittent theta burst stimulation (iTBS) is a novel protocol that consists of intermittently delivering bursts of 3 TMS pulses at high frequency (50 Hz) every 200 ms for 2 s (5Hz) every 10 s (total 600 pulses), allowing for greater long-lasting effects on cortical excitability and a more important number of rTMS pulses to be delivered in a shorter duration than standardized high frequency (HF) rTMS protocols. iTBS induces a long-term potentiation (LTP)-like effect by increasing the postsynaptic concentration of calcium ions and has been applied to treat MDD. iTBS has been proved to be safe and well tolerated and to have antidepressant properties. Prolonged iTBS (piTBS, total 1800 pulses) has been recently applied to treat MDD with favorable antidepressant properties. An accelerated protocol of piTBS has been recently approved to treat medication-refractory MDD by FDA.

MDD is associated with a 2.3 fold increase in prevalence of suicidal ideation as compared to the general population. The lifetime rate of death due to suicide among MDD patients is 15-20%. Research indicates that 30% of TRD patients will attempt suicide during their lifetime, which is a two-to-four times greater proportion than MDD patients who respond to treatment. Research indicates that rTMS improves several preconditions for suicide, including mood, memory, attention, executive functioning. rTMS is thought to have molecular effects similar to those seen with electroconvulsive therapy (ECT), which is effective in treating suicidal patients, such as increased BDNF, increased monoamine turnover and normalization of the hypothalamic-pituitary-adrenal axis. Some research indicates that rTMS may reduce suicidal ideations of patients with MDD. However, powered sham-controlled rTMS clinical trials focusing on the efficacy to improve suicide risks are limited.

The study aims to investigate the efficacy of accelerated piTBS over the left DLPFC as an add-on therapy to improve suicide ideations in TRD patients. Moreover, it provides data on other secondary outcomes and neurophysiological data for this intervention condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 20-65 years, met criteria for DSM-V major depressive disorder.
* A depression severity score of 18 or more on the 17-item Hamilton Rating Scale for Depression (HRSD-17) as well as a score of 1 or more on the item of the HDRS-17 (item 3).
* Meeting criteria for TRD defined as no clinical response to at least one adequate trial of one major class of antidepressants.
* Having been receiving stable antidepressant medications regimen for more than 4 weeks before enrollment and having their original medication regimen unchanged throughout the trial.

Exclusion Criteria:

* Having MDD with psychotic features, bipolar disorder, schizophrenia, organic brain syndrome or active substance (except for tobacco and coffeine) use disorder.
* Having previous intracranial surgery and ferromagnetic metallic implants in the head.
* History of brain abnormalities (e.g., brain neoplasms, arteriovenous malformations, meningitis, encephalitis, epilepsy, neurodegenerative disorders).
* Pregnancy at enrollment.
* History of treatment with electroconvulsive therapy (ECT) or no response to rTMS over the left DLPFC.
* Those who had attempted a suicide within six months from the screening date.
* Skin lesions on scalp at the area of coil application.
* In addition to those listed above, those who were deemed unsuitable for participating in this clinical trial by the medical judgment of the investigator due to other reasons (e.g., lack of competence to consent to research or any other contraindications to receiving rTMS).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
The change over time in the score of Beck Scale for Suicide Ideation (BSS) (from baseline to the timepoints at 1 week after piTBS, at the end of piTBS, and at 1, 2, and 4 weeks after piTBS). | 6 weeks
  BSS is a 21-item self-report instrument for detecting and measuring the current intensity of the patients' specific attitudes, behaviors, and plans to commit suicide during the past week.

SECONDARY OUTCOMES:
The change over time in the score of Snaith-Hamilton Pleasure Scale (SHAPS) (from baseline to the timepoints at 1 week after piTBS, at the end of piTBS, and at 1, 2, and 4 weeks after piTBS). | 6 weeks
  SHAPS is a 14-item self-report questionnaire to assess subject's pleasure experience in the "last few days". It is rated from definitely agree to definitely disagree on a 4-point Likert scale (i.e., scoring from 1 to 4) and the total score ranges from 14 to 56. Higher scores indicate more severe anhedonia.
The change over time in the score of Beck Hopelessness Scale (BHS) (from baseline to the timepoints at 1 week after piTBS, at the end of piTBS, and at 1, 2, and 4 weeks after piTBS). | 6 weeks
  BHS is 20-item questionnaire measuring pessimism/hopelessness, a construct related to suicide ideations.
The change over time in the score of Montgomery-Å sberg Depression Rating Scale (MADRS) (from baseline to the timepoints at 1 week after piTBS, at the end of piTBS, and at 1, 2, and 4 weeks after piTBS). | 6 weeks
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item tool to measure the severity of depressive episodes. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
The change over time in the score of 17-item Hamilton Depression Rating Scale (HDRS) (from baseline to the timepoints at 1 week after piTBS, at the end of piTBS, and at 1, 2, and 4 weeks after piTBS). | 6 weeks
  The Hamilton Rating Scale for Depression is a 17-item instrument that was designed to measure frequency and intensity of depressive symptoms in individuals with major depressive disorder. Ratings are made using either a five- or a three-point scale, yielding total scores from 0 to 61.
The change over time in the score of Hamilton Anxiety Rating Scale (HAM-A) (from baseline to the timepoints at 1 week after piTBS, at the end of piTBS, and at 1, 2, and 4 weeks after piTBS). | 6 weeks
  The HAM-A was to measure the severity of anxiety symptoms, consisting of 14 items, each defined by a series of symptoms, and measures both psychic anxiety and somatic anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56.
The change over time in the score of Young Mania Rating Scale (YMRS) (from baseline to the timepoints at 1 week after piTBS, at the end of piTBS, and at 1, 2, and 4 weeks after piTBS). | 6 weeks
  The YMRS is a scale to assess manic symptoms. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale.
The changes over time in the results of Wisconsin Card Sorting Test (WCST) (from baseline to the timepoint at the end of piTBS). | 2 weeks
  A neuropsychological test of "set-shifting", i.e. the ability to display flexibility in the face of changing schedules of reinforcement.
The changes over time in the results of Color Trails Test (CTT) (from baseline to the timepoint at the end of piTBS). | 2 weeks
  The CTT, a culture-neutral version of the Trail Making Test, was selected to measure sustained visual attention. The CTT consists of two parts (CTT-1 and CTT-2). The CTT-1 requires participants to connect a series of numbered circles that are randomly printed on a sheet of paper. In the CTT-2, numbered circles of 1 to 25 are shown twice (printed in pink and in yellow) randomly on a sheet of paper. Participants are asked to connect the numbers from 1 to 25 alternating between the two colors.
The changes over time in the results of Stroop Color Word Test (SCWT) (from baseline to the timepoint at the end of piTBS). | 2 weeks
  Stroop Color Word Test (SCWT), Chinese version; was administered to measure selective attention and cognitive flexibility. SCWT is composed of three parts, each lasting for 45 seconds.
The changes over time in the results of indices of heart rate variability (HRV) (from baseline to the timepoint at the end of piTBS) and the HRV indices during each piTBS session. | 2 weeks
  HRV indices represent autonomic functioning. ECG electrodes were placed on bilateral arms just below the elbows, with a ground electrode placed just above the right wrist bone. For HRV indices measured at baseline and the end of piTBS, lead I electrocardiogram of each patient was taken for 5 min after sitting and having a rest for 20 min in a soundproof, dim-lighted room with thermostatic control. For HRV indices measured during each piTBS session, lead I electrocardiogram of each patient was taken for 11 min. The ECG signals were acquired, stored, pre-processed according to the recommended procedures and processed by an HRV analyser. The time domain of HRV is obtained: Standard deviation of NN intervals (SDNN). Power spectrum of HRV is quantified into the standard frequency-domain measurements including low-frequency power (LF, 0.04-0.15 Hz), high-frequency power (HF, 0.15- 0.40 Hz).
The changes over time in EEG absolute power and lag phase synchronization in the frontal electrodes in the delta, theta, alpha, beta and gamma range (from baseline to the end of piTBS). | 2 weeks
  In a recliner in a dimly lit, electrically shielded room, patients' EEGs were recorded at baseline and at the end of piTBS by using the full-band DC-EEG system with 32 EEG Ag/AgCl electrodes in the extended 10-20 International placement. EEG will be collected with eye opened (5min) and closed (5min). Signals will be amplified in the dynamic input range of ± 140 mV at a resolution of 0.5 μV by using EEG amplifiers and stored for offline analyses. Eye or muscle artifacts were automatically detected and removed.
The changes over time in high density near infrared spectroscopy (from baseline to the end of piTBS). | 2 weeks
  Resting-state and cognitive-task protocol used for the functional near infrared spectroscopy (fNIRS) system to measure the relative changes in oxy Hb. Hemoglobin Hb changes will be measured during a resting state (for 3 min) and 2 different cognitive tasks (each for around 5 min): semantic verbal fluency task (SVFT) and a 2 back task. An SVFT involves generating as many words as possible within a certain time frame and hints at the semantic category of the words generated. The 2 back task is used to evaluate participants' working memory.
The changes over time in the results of Digit Symbol Substitution Test (DSST) (from baseline to the timepoint at the end of piTBS). | 2 weeks
  The Digit Symbol Substitution Test (DSST) is a performance-based test of cognitive performance tapping into processing speed, executive function, and attention. It has a 90-s test period and a score range from 0 to 133.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-An Chang, MD, Principal Investigator — Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan
Locations (1):
- Tri-service general hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No